CLINICAL TRIAL: NCT04274439
Title: Effectiveness and Cost-Effectiveness of a Tele-Rehabilitation Program in the Treatment of Chronic Musculoskeletal Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Cidade de Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Dr Bruno Saragiotto, Assistant Professor, Universidade Cidade de Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 02892918.0.0000.8084; 2016/24217-7 (Other Grant/Funding Number: FAPESP (São Paulo Research Foundation))
Record Dates: First submitted 2019-05-09; First posted 2020-02-18 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Chronic Pain
Keywords: Chronic Pain; Telerehabilitation; Telemedicine; Physical Therapy
MeSH Terms: conditions — Chronic Pain | interventions — Exercise; Telerehabilitation

STUDY DESIGN:
Intervention Model Description: This is a controlled clinical trial, with the Intervention group performing the 8-week follow-up and access to 8 pain education videos and 8 exercise videos prescribed for patients with chronic pain, and the control group receiving information on chronic pain for one booklet. Randomized through site programming, so that the subject enters his / her login and password and is directed to one of the study groups, with blind evaluator without access to randomization information throughout the course of the study and follow-up of the outcome measures for 3 , 6 and 12 months after randomization.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet-Based Pain Education and Exercise (Experimental): Patients allocated to the intervention group will receive a login and password for individual access to the website designed for the study. The content of this intervention will include videos and animations based on pain education, physical activity promotion and general exercises. The pain education component will be based on the E-pain intervention developed by Reis et al (2017), which includes nine main features: (1) acceptance, (2 and 3) education about pain, (4) sleep hygiene, (5) recognizing stress and negative emotions, (6) increasing positive coping in lifestyle, (7) exercises, (8) communication and (9) relapse prevention. The exercise component will include general exercises aiming to improve strength, flexibility, control and coordination.
  Patients in this group will also receive weekly text messages and a health coaching over the telephone. The text messages will include information on the benefits of exercises, motivation, and positive messages about dealing with pain.
  Interventions: Other: Internet-Based Pain Education and Exercise
- Online Booklet (Active Comparator): The patients allocated to the control group will have access to an online booklet containing general information about self-management of chronic pain, including pain education, advice on healthy lifestyle and sleeping habits and promotion of exercises. They will also receive one phone call at week 4 and text messages once a week during the study period.
  Interventions: Other: Online Booklet

INTERVENTIONS:
Other: Internet-Based Pain Education and Exercise — Telerehabilitation is defined as providing techniques for therapeutic rehabilitation remotely or off-site using telecommunication technologies. Thus, our intervention will be based on the use of a website created and registered especially for the study that will have the shooting of 1 video of pain education and 1 video of exercises for the subjects of the study, totaling 8 videos of pain education and 8 exercise videos. We will provide complimentary materials along with the triggered videos and a booklet of chronic pain information. We will also make weekly calls for a health coaching service and the sending of smartphone messages for the motivation and accountability of the subjects.
  Other Names: Telerehabilitation
  Arms: Internet-Based Pain Education and Exercise
Other: Online Booklet — An online booklet containing information about chronic pain and suggestions for lifestyle modifications and behavior will be delivered, as well as an incentive to perform physical exercises.
  Arms: Online Booklet

SUMMARY:
The aim of this clinical trial is to develop and test the effectiveness and cost-effectiveness of an internet-based self-management program based on pain education and exercise for people with chronic musculoskeletal pain.

DETAILED DESCRIPTION:
Chronic pain is a major burden on the individual and society. It is estimated that about one third of the adult population worldwide suffer from chronic pain, with higher prevalence rates reported for low-income countries. Internet-based self-management programs have grown with the development of new technologies and have been extensively used for delivering healthcare in many areas. However, there is still little research on the development and testing of remotely-delivered programs for the management of chronic musculoskeletal pain, especially in low and mid-income countries. The aim of this clinical trial is to develop and test the effectiveness and cost-effectiveness of an internet-based self-management program based on pain education and exercise for people with chronic musculoskeletal pain.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 60 years
* Seeking treatment for any chronic musculoskeletal pain of at least 3 points in a 0 to 10 Pain Numerical Rating Scale
* Able to read and understand Portuguese
* With internet access.

  * Chronic Pain will be defined as pain lasting more than 12 weeks.

Exclusion Criteria:

* Present neurological symptoms (nerve root compromise, or sensation deficits)
* Present serious spinal pathologies (e.g., fracture, tumor, inflammatory, autoimmune, and infectious diseases)
* Present serious cardiovascular and metabolic diseases (e.g., coronary heart disease, cardiac insufficiency, decompensated diabetes)
* Recent orthopaedic surgery (over the last 12 months)
* Scheduled to undergo surgery in the next 6 months, or pregnancy
* If have any contraindication to exercise

  * We will perform a pre-screening for physical activity participation at baseline using the Physical Activity Readiness Questionnaire (PAR-Q) Portuguese version to rule out any contraindication to participate in physical activity.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2020-03-03 (Actual); Primary Completion 2021-09-02 (Estimated); Study Completion 2022-03-10 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity at post-treatment follow-up | Post-treatment follow-up (8 weeks)
  The primary outcome will be pain intensity measured using the Pain Numerical Rating Scale, a numerical scale of 11 domains, where 0 indicates no pain and 10 indicates maximum pain intensity.

SECONDARY OUTCOMES:
Pain intensity at 6 months and 12 months follow-up | 6 months and 12 months follow-up
  TMeasured using the Pain Numerical Rating Scale, a numerical scale of 11 domains, where 0 indicates no pain and 10 indicates maximum pain intensity.
Function | The outcome will be evaluated after the treatment period (8 weeks), after 6 months of randomization and after 12 months of randomization of each subject.
  Measured with the Patient Specific Functional Scale, a self-reported scale specific for the measurement of functionality in musculoskeletal injuries, where the patient classifies his activities from 0 to 10, being 0 the inability to perform that function and 10 the total capacity to perform the function;
Health-Related Quality of Life | The outcome will be evaluated after the treatment period (8 weeks), after 6 months of randomization and after 12 months of randomization of each subject.
  Measured with the SF-12, a self-reported questionnaire with 12 questions and classification of 8 different dimensions related to quality of life. Higher scores define better quality of life;
Kinesiophobia | The outcome will be evaluated after the treatment period (8 weeks), after 6 months of randomization and after 12 months of randomization of each subject.
  Measured with the Tampa Scale of Kinesiophobia, a self-reported questionnaire with 17 questions, where the patient ranks "totally disagree" statements equivalent to one point, "partially disagree", two points, "partially agree", three points and "totally agree", four points . Higher scores at the end of the questionnaire identify worse results in kinesiophobia outcome;
Global Perceived Effect | The outcome will be evaluated after the treatment period (8 weeks), after 6 months of randomization and after 12 months of randomization of each subject.
  Measured with the Global Perceived Effect Scale, a self-reported scale, with scores of -5 to 5, where the progression of the patient's condition will be classified from a certain point in time. Scores of -5 indicate a lot of worsening and scores of 5 indicate a lot of improvement.
Anxiety and Depression | The outcome will be evaluated after the treatment period (8 weeks), after 6 months of randomization and after 12 months of randomization of each subject.
  Measured by the Hospital Anxiety and Depression Scale, a self-reported scale with 14 questions, 7 for depression and 7 for anxiety. Each question has a rating ranging from 0 to 3 according to the patient's response. Scores near 21 indicate the worst results.
Pain Catastrophisation | The outcome will be evaluated after the treatment period (8 weeks), after 6 months of randomization and after 12 months of randomization of each subject.
  Measured with the Pain Catastrophising Scale, a self-reported scale with 13 statements, where the patient ranks the affirmations between 0 being "minimal" to 4 "very intense." The calculation of the final score is based on 3 subdomains of the scale and scores closer to 52 indicate worse results.
Pain-related Attitudes and Beliefs | The outcome will be evaluated after the treatment period (8 weeks), after 6 months of randomization and after 12 months of randomization of each subject.
  Measured with Orebro Musculoskeletal Pain Questionnaire, a self-reported questionnaire with questions related to musculoskeletal pain classified from 0 to 10 and its score calculated later according to these answers and using an own algorithm of the questionnaire.
Self-efficacy | The outcome will be evaluated after the treatment period (8 weeks), after 6 months of randomization and after 12 months of randomization of each subject.
  Measured with Pain Self-Efficacy Questionnaire, a questionnaire with 22 questions classified in three domains, with a score of each domain ranging from 10 to 100. A total score close to 300 indicates a greater sense of self-efficacy.
Adverse Effects | The outcome will be evaluated after the treatment period (8 weeks), after 6 months of randomization and after 12 months of randomization of each subject.
  Measured by recording the number of adverse events during the intervention period.

OTHER OUTCOMES:
Patient's Expectancy for Improvement at Baseline | The outcome will be evaluated at the baseline
  Expectancy of Improvement Numerical Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno T Saragiotto, PostDoc, Principal Investigator — Universidade Cidade de Sao Paulo
Locations (1):
- Rua Cesário Galeno, 448/475, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
We can share our data upon request.

REFERENCES:
- [Background] Elzahaf RA, Tashani OA, Unsworth BA, Johnson MI. The prevalence of chronic pain with an analysis of countries with a Human Development Index less than 0.9: a systematic review without meta-analysis. Curr Med Res Opin. 2012 Jul;28(7):1221-9. doi: 10.1185/03007995.2012.703132. Epub 2012 Jul 2. PMID 22697274
- [Background] Fayaz A, Croft P, Langford RM, Donaldson LJ, Jones GT. Prevalence of chronic pain in the UK: a systematic review and meta-analysis of population studies. BMJ Open. 2016 Jun 20;6(6):e010364. doi: 10.1136/bmjopen-2015-010364. PMID 27324708
- [Background] Global Burden of Disease Study 2013 Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 301 acute and chronic diseases and injuries in 188 countries, 1990-2013: a systematic analysis for the Global Burden of Disease Study 2013. Lancet. 2015 Aug 22;386(9995):743-800. doi: 10.1016/S0140-6736(15)60692-4. Epub 2015 Jun 7. PMID 26063472
- [Background] Chen B, Li L, Donovan C, Gao Y, Ali G, Jiang Y, Xu T, Shan G, Sun W. Prevalence and characteristics of chronic body pain in China: a national study. Springerplus. 2016 Jun 30;5(1):938. doi: 10.1186/s40064-016-2581-y. eCollection 2016. PMID 27386382
- [Background] Park PW, Dryer RD, Hegeman-Dingle R, Mardekian J, Zlateva G, Wolff GG, Lamerato LE. Cost Burden of Chronic Pain Patients in a Large Integrated Delivery System in the United States. Pain Pract. 2016 Nov;16(8):1001-1011. doi: 10.1111/papr.12357. Epub 2015 Oct 7. PMID 26443292
- [Background] Woby SR, Roach NK, Urmston M, Watson PJ. The relation between cognitive factors and levels of pain and disability in chronic low back pain patients presenting for physiotherapy. Eur J Pain. 2007 Nov;11(8):869-77. doi: 10.1016/j.ejpain.2007.01.005. Epub 2007 Mar 13. PMID 17360202
- [Background] Woby SR, Urmston M, Watson PJ. Self-efficacy mediates the relation between pain-related fear and outcome in chronic low back pain patients. Eur J Pain. 2007 Oct;11(7):711-8. doi: 10.1016/j.ejpain.2006.10.009. Epub 2007 Jan 10. PMID 17218132
- [Background] Foster NE, Thomas E, Bishop A, Dunn KM, Main CJ. Distinctiveness of psychological obstacles to recovery in low back pain patients in primary care. Pain. 2010 Mar;148(3):398-406. doi: 10.1016/j.pain.2009.11.002. Epub 2009 Dec 22. PMID 20022697
- [Background] Truchon M. Determinants of chronic disability related to low back pain: towards an integrative biopsychosocial model. Disabil Rehabil. 2001 Nov 20;23(17):758-67. doi: 10.1080/09638280110061744. PMID 11762878
- [Background] Lotze M, Moseley GL. Theoretical Considerations for Chronic Pain Rehabilitation. Phys Ther. 2015 Sep;95(9):1316-20. doi: 10.2522/ptj.20140581. Epub 2015 Apr 16. PMID 25882484
- [Background] Ballantyne JC, Sullivan MD. Intensity of Chronic Pain--The Wrong Metric? N Engl J Med. 2015 Nov 26;373(22):2098-9. doi: 10.1056/NEJMp1507136. No abstract available. PMID 26605926
- [Background] Dear BF, Titov N, Perry KN, Johnston L, Wootton BM, Terides MD, Rapee RM, Hudson JL. The Pain Course: a randomised controlled trial of a clinician-guided Internet-delivered cognitive behaviour therapy program for managing chronic pain and emotional well-being. Pain. 2013 Jun;154(6):942-50. doi: 10.1016/j.pain.2013.03.005. PMID 23688830
- [Background] Lundell S, Holmner A, Rehn B, Nyberg A, Wadell K. Telehealthcare in COPD: a systematic review and meta-analysis on physical outcomes and dyspnea. Respir Med. 2015 Jan;109(1):11-26. doi: 10.1016/j.rmed.2014.10.008. Epub 2014 Oct 27. PMID 25464906
- [Background] Cottrell MA, Galea OA, O'Leary SP, Hill AJ, Russell TG. Real-time telerehabilitation for the treatment of musculoskeletal conditions is effective and comparable to standard practice: a systematic review and meta-analysis. Clin Rehabil. 2017 May;31(5):625-638. doi: 10.1177/0269215516645148. Epub 2016 May 2. PMID 27141087
- [Background] Khan F, Amatya B, Kesselring J, Galea MP. Telerehabilitation for persons with multiple sclerosis. A Cochrane review. Eur J Phys Rehabil Med. 2015 Jun;51(3):311-25. Epub 2015 May 6. PMID 25943744
- [Background] de Boer MJ, Versteegen GJ, Vermeulen KM, Sanderman R, Struys MM. A randomized controlled trial of an Internet-based cognitive-behavioural intervention for non-specific chronic pain: an effectiveness and cost-effectiveness study. Eur J Pain. 2014 Nov;18(10):1440-51. doi: 10.1002/ejp.509. Epub 2014 Apr 29. PMID 24777973
- [Background] Cryer L, Shannon SB, Van Amsterdam M, Leff B. Costs for 'hospital at home' patients were 19 percent lower, with equal or better outcomes compared to similar inpatients. Health Aff (Millwood). 2012 Jun;31(6):1237-43. doi: 10.1377/hlthaff.2011.1132. PMID 22665835
- [Background] Costa LO, Maher CG, Latimer J, Ferreira PH, Ferreira ML, Pozzi GC, Freitas LM. Clinimetric testing of three self-report outcome measures for low back pain patients in Brazil: which one is the best? Spine (Phila Pa 1976). 2008 Oct 15;33(22):2459-63. doi: 10.1097/BRS.0b013e3181849dbe. PMID 18923324
- [Background] Reis FJJ, Bengaly AGC, Valentim JCP, Santos LC, Martins EF, O'Keeffe M, Meziat-Filho N, Nogueira LC. An E-Pain intervention to spread modern pain education in Brazil. Braz J Phys Ther. 2017 Sep-Oct;21(5):305-306. doi: 10.1016/j.bjpt.2017.06.020. Epub 2017 Aug 19. No abstract available. PMID 28864352
- [Derived] Fioratti I, Miyamoto GC, Fandim JV, Ribeiro CPP, Batista GD, Freitas GE, Palomo AS, Reis FJJD, Costa LOP, Maher CG, Saragiotto BT. Feasibility, Usability, and Implementation Context of an Internet-Based Pain Education and Exercise Program for Chronic Musculoskeletal Pain: Pilot Trial of the ReabilitaDOR Program. JMIR Form Res. 2022 Aug 30;6(8):e35743. doi: 10.2196/35743. PMID 35776863
- [Derived] Fioratti I, Saragiotto BT, Reis FJJ, Miyamoto GC, Lee H, Yamato TP, Fandim JV, Dear B, Maher CG, Costa LOP. Evaluation of the efficacy of an internet-based pain education and exercise program for chronic musculoskeletal pain in comparison with online self-management booklet: a protocol of a randomised controlled trial with assessor-blinded, 12-month follow-up, and economic evaluation. BMC Musculoskelet Disord. 2020 Jun 26;21(1):404. doi: 10.1186/s12891-020-03423-x. PMID 32590959